CLINICAL TRIAL: NCT04209582
Title: Transcutaneous Oxygen Pressure of the Injured Ankle as Predictor of Postoperative Cutaneous Pain
Acronym: TAC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0303
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: measurement of TcPO2 with skin electrode — measurement of TcPO2 with skin electrode

SUMMARY:
This monocentric prospective observational pilot study aims to investigate if the measurement of TcPO2 can be used as a predictor of postoperative cutaneous pain in patients with ankle surgery.

DETAILED DESCRIPTION:
This prospective observational study aims to determine the limit of TcPO2 predictive of postoperative cutaneous pain in patients with ankle trauma.

A TcPO2 measurement will be performed preoperatively at the patient's arrival in the emergency room, then every day after the operation for 3 days and finally at the follow-up visits at 3 and 6 weeks.

The cutaneous pain is evaluated by a PSAS self-questionnaire (completed by the patient) and an OSAS questionnaire (completed by the surgeon). These grids evaluate the tolerance and cicatricial quality in the medium and long term by the operator and the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgery of ankle trauma

Exclusion Criteria:

* Patient who does not agree to participate
* Patient unable to express agreement (ex: unconscious)
* Minor patient
* Major patient under tutorship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population studied concerns all adult patients suffering from ankle trauma requiring surgical management, it is heterogeneous, concerns all ages, regardless of co-morbidities. Minor patients and patients unable to give their consent will not be included.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Presence of postoperative skin pain within 3 months postoperatively | 0-3 Month

SECONDARY OUTCOMES:
Preoperative TcPO2 on the injured ankle and contralateral ankle | day 0
  compare TcPO2 values between healthy ankle and traumatized ankle
Preoperative and postoperative day 1 TcPO2 on the injured ankle | Day 1
  Compare TcPO2 values before and after surgery
Rates of postoperative complications related to S12 surgery and TcPO2 measurements | 3 months
  Measure surgical complications based on TcPo2 measurements
Surgical revision rate at S12 and TcPO2 measurements | 3 months
  Measure the number of surgical revisions based on TcPo2 measurements
Preoperative and postoperative day 1 TcPO2 on the injured ankle and type of fracture | Day 1
  Describe the TcPO2 measurements according to the type of fracture
Preoperative and postoperative day 1 TcPO2 on the injured ankle and comorbidities such as pulmonary pathologies, microangiopathy, vascular pathologies, history of trauma | Day 1
  Describe the measures of TcPO2 according to comorbidities
Patient scar assessment scale (PSAS grid) at S6 and S12 | Week 6
  Describe the type of skin pain according to TcPO2 measurement The PSAS observation scale consists of 7 questions for the patient concerning pain, itching, colour, suppleness, thickness, appearance and a general opinion on the scar.
  Each parameter is rated on a scale from 1 (best score) to 10 (worst score). The sum of the 7 parameters gives the total score (minimum value = 7 ; maximum value = 70).
Patient scar assessment scale (PSAS grid) at S6 and S12 | Week 12
  Describe the type of skin pain according to TcPO2 measurement The PSAS observation scale consists of 7 questions for the patient concerning pain, itching, colour, suppleness, thickness, appearance and a general opinion on the scar.
  Each parameter is rated on a scale from 1 (best score) to 10 (worst score). The sum of the 7 parameters gives the total score (minimum value = 7 ; maximum value = 70).
OSAS Scale (observer scars assessment scale) at S6 and S12 | Week 6
  Measure the quality of healing The OSAS observation scale consists of seven parameters (vascularization, pigmentation, thickness, relief, plasticity, surface and a global evaluation).
  Each parameter is rated on a scale ranging from 1 ("like normal skin") to 10 ("the worst scar imaginable").
  The sum of the 7 parameters gives the observer's total score (minimum value = 7 ; maximum value = 70).
OSAS Scale (observer scars assessment scale) at S6 and S12 | Week 12
  Measure the quality of healing The OSAS observation scale consists of seven parameters (vascularization, pigmentation, thickness, relief, plasticity, surface and a global evaluation).
  Each parameter is rated on a scale ranging from 1 ("like normal skin") to 10 ("the worst scar imaginable").
  The sum of the 7 parameters gives the observer's total score (minimum value = 7 ; maximum value = 70).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Brulefert, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided